CLINICAL TRIAL: NCT02500303
Title: Rehabilitation & Function Following Lower Limb Amputation: the Influence of Diabetes
Brief Title: Influence of Diabetes on Lower Limb Amputation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Glasgow (Other)
Collaborators: NHS Greater Glasgow and Clyde Board HQ (Other)
Responsible Party: Principal Investigator, Fiona Smith, PhD Student & Chief Investigator, University of Glasgow
Other Study IDs: GN13DI563
Record Dates: First submitted 2014-12-02; First posted 2015-07-16 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Diabetes; PAD
Keywords: Amputation
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to explore the factors that influence limb fitting in those with diabetes compared to those without diabetes. The population without diabetes will usually present with peripheral arterial disease (PAD) and are similar in management following LEA. The impact that not walking with a prosthesis has long term on both populations will be explored. In general, previous research has used retrospective analysis of case notes which, although valuable, have fixed fields and only allow the researcher to look at associations between factors not at causation. Additionally, very few have followed a population over time. Therefore this study will be a prospective observational analysis of all those who undergo a LEA in one year from 01/03/14 to 28/02/15 within the Greater Glasgow & Clyde area with follow up at 6, 12 & 18 months from date of amputation.

DETAILED DESCRIPTION:
This research has been designed to ask the following question: What are the factors that influence the rehabilitation and functional outcomes following LEA, in the long term in both those with and without diabetes.

Therefore this study will be a prospective observational analysis of all those who undergo a LEA in one year within the Greater Glasgow & Clyde area with follow up at 6, 12 & 18 months from date of amputation.

* Primary Endpoint Comparison of rehabilitation and functional outcomes in those with diabetes to those without diabetes, up to 18 months post LEA.
* Secondary endpoints

  1. At discharge from rehabilitation, the characteristics of those who proceed to limb fitting following LEA to those who do not will be defined.
  2. At discharge from rehabilitation, the characteristics of those with diabetes that do not proceed to limb fitting following LEA compared to those who do.
  3. At discharge from rehabilitation to 18 months post LEA, a comparison of the characteristics in those with and without diabetes.
  4. From six months post LEA, at 6 monthly intervals (6,12 & 18 months), a comparison of the health status, social circumstances, mobility and quality of life measures in those with and without diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age with a major amputation above the ankle.

Exclusion Criteria:

* Amputation for tumour, trauma, congenital abnormalities
* Amputation at hip disarticulation or trans-pelvectomy level
* Adults with incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All persons over 18 years old undergoing a lower limb amputation for Diabetes and / or peripheral arterial disease within the Greater Glasgow & Clyde area.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 3 years
  Date of Death if applicable
Limb fitting | 3 years
  Dtae of receiving prosthetic limb
Length of stay | 3 years
  Length of time in hospital as an in patient
Readmission | 3 years
  Date of readmission to hospital
Further surgery | 3 years
  Number and level of further amputations

SECONDARY OUTCOMES:
EQ-5D-5L | 3 years
  Quality of life measure
Reintegration to normal living index | 3 years
Prosthetic Limb User Mobility | 3 years
  As assessed by the prosthetic limb user survey mobility scale
Co-morbidities | 3 years
  Functional co-morbidity index

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Paul, PhD, Study Director — University of Glasgow
Locations (1):
- Western Infirmary, Glasgow, United Kingdom